CLINICAL TRIAL: NCT01444456
Title: Electronic Assessment of Quality of Life in Patients With Symptomatic Chemotherapy-induced Anaemia: An International Prospective Observational Study (eAQUA)
Brief Title: Assessment of Quality of Life in Patients With Symptomatic Chemotherapy-induced Anaemia
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101123
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Anemia; Breast Cancer; Cancer; Colorectal Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Solid Tumors; Bladder Cancer; Endometrial Cancer; Renal Cancer; Pancreatic Cancer; Esophageal Cancer; Gastric Cancer
Keywords: Breast Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Colorectal Cancer; Aranesp; Chemotherapy induced anaemia; Chemotherapy; Bladder Cancer; Endometrial Cancer; Renal Cancer; Pancreatic Cancer; Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Anemia; Breast Neoplasms; Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Endometrial Neoplasms; Kidney Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Darbepoetin alfa: Participants receiving systemic chemotherapy for solid tumors who also received darbepoetin alfa (Aranesp®) to treat symptomatic anemia according to routine institutional practice.
- Cohort 2: Any ESA: Participants receiving systemic chemotherapy for solid tumors who also received darbepoetin alfa (Aranesp®) or another erythropoiesis-stimulating agent (ESA) to treat symptomatic anemia according to routine institutional practice.

SUMMARY:
This is a multicenter, international, prospective, observational study of patients who are receiving systemic chemotherapy for solid tumour cancers (breast, colorectal, ovarian, prostate, lung, bladder, endometrial, renal, pancreatic, esophageal or gastric) and who are receiving darbepoetin alfa (Aranesp®) or other erythropoiesis-stimulating agent (ESA) to treat symptomatic anaemia.

Quality of Life will be assessed electronically with the aim of estimating improvement in quality of life for those patients receiving darbepoetin alfa (Aranesp®) who also have an increase in haemoglobin (Hb) of ≥1 g/dL

DETAILED DESCRIPTION:
Before enrolling participants, each country was assigned to either cohort 1 (patients receiving only darbepoetin alfa) or cohort 2 (patients receiving any ESA). Cohort 2 was assigned only to those countries in which local regulations did not permit observational study participation by patients receiving a specific agent in a drug class.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast, colorectal, ovarian, prostate, lung, bladder, endometrial, renal, pancreatic, esophageal or gastric cancer
* Expected to receive at least 8 additional weeks of a given regimen of myelosuppressive chemotherapy after enrolment
* Starting treatment with either darbepoetin alfa (in Cohort 1 countries) or any ESA (in Cohort 2 countries) as per European Summary of Product Characteristics (SPC) for symptomatic anaemia.

Exclusion Criteria:

* Received any ESA treatment or Red Blood Cell (RBC) transfusion within 28 days prior to enrolment
* Known primary benign or malignant haematologic disorder which can cause anaemia
* Known hypersensitivity to ESAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with either breast, colorectal, ovarian, prostate, lung, bladder, endometrial, renal, pancreatic, esophageal or gastric cancer who will receive darbepoetin alfa (Aranesp®) or other erythropoiesis-stimulating agent (ESA) for the treatment of symptomatic chemotherapy-induced anaemia (CIA) in routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 1262 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (104):
- Austria (6):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Vöcklabruck
  - Research Site, Wels
- Belgium (11):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Eupen
  - Research Site, Gilly
  - Research Site, Mechelen
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Sint-Niklaas
  - Research Site, Verviers
- France (37):
  - Research Site, Aix-en-Provence
  - Research Site, Amiens
  - Research Site, Aubagne
  - Research Site, Bayonne
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Boulogne Sur Mer Cédex
  - Research Site, Bourg-en-Bresse
  - Research Site, Brive-la-Gaillarde
  - Research Site, Carcassonne
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Dijon
  - Research Site, Draguignan
  - Research Site, La Seyne-sur-Mer
  - Research Site, Le Mans
  - Research Site, Longjumeau
  - Research Site, Marseille
  - Research Site, Mont-de-Marsan
  - Research Site, Montauban
  - Research Site, Nancy
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Périgueux
  - Research Site, Pontoise
  - Research Site, Pringy
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Quentin
  - Research Site, Soissons
  - Research Site, Soyaux
  - Research Site, Strasbourg
  - Research Site, Vichy
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Bremerhaven
  - Research Site, Cologne
  - Research Site, Gelsenkirchen
  - Research Site, Goslar
  - Research Site, Halle
  - Research Site, Mannheim
  - Research Site, Neunkirchen
  - Research Site, Rotenburg (Wümme)
  - Research Site, Soest
  - Research Site, Stralsund
  - Research Site, Würselen
- Greece (4):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Marousi
  - Research Site, Papagou
- Italy (5):
  - Research Site, Cefalù PA
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Torino
- Netherlands (8):
  - Research Site, Amstelveen
  - Research Site, Dordrecht
  - Research Site, Enschede
  - Research Site, Flushing
  - Research Site, Leiderdorp
  - Research Site, Purmerend
  - Research Site, Roosendaal
  - Research Site, Zutphen
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Konin
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lubin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wroclaw
- Romania (9):
  - Research Site, Alba Iulia
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Oradea
  - Research Site, Râmnicu Vâlcea
  - Research Site, Târgu Mureş
  - Research Site, Timișoara

REFERENCES:
- [Background] Mouysset JL, Freier B, van den Bosch J, Levache CB, Bols A, Tessen HW, Belton L, Bohac GC, Terwey JH, Tonini G. Hemoglobin levels and quality of life in patients with symptomatic chemotherapy-induced anemia: the eAQUA study. Cancer Manag Res. 2016 Jan 21;8:1-10. doi: 10.2147/CMAR.S88110. eCollection 2016. PMID 26855598
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open to patients receiving systemic chemotherapy for solid tumors who also received darbepoetin alfa or another erythropoiesis-stimulating agent (ESA) to treat symptomatic anemia. First patient enrolled 10 october 2011; last patient enrolled 28 May 2013.
Pre-assignment Details: Before enrolling participants, each country was assigned to either cohort 1 (patients receiving only darbepoetin alfa) or cohort 2 (patients receiving any ESA). Cohort 2 was assigned only to those countries in which local regulations did not permit observational study participation by participants receiving a specific agent in a drug class.
Groups:
- Darbepoetin Alfa or Other ESA: Participants receiving systemic chemotherapy for solid tumors who also received darbepoetin alfa (Aranesp®) or another erythropoiesis-stimulating agent (ESA) to treat symptomatic anemia according to routine institutional practice.
Period: Overall Study
Arm/Group | Darbepoetin Alfa or Other ESA
Started | 1262
Received Darbepoetin Alfa or Other ESA | 1158
Received Darbepoetin Alfa | 1134
Completed | 977 (Defined as 4 weeks after last dose of ESA or chemotherapy or 13 weeks after enrolment)
Not Completed | 285
Not completed — Withdrawal by Subject | 21
Not completed — Physician Decision | 9
Not completed — Lost to Follow-up | 37
Not completed — Death | 73
Not completed — Ineligibility determined | 23
Not completed — Other | 18
Not completed — Not treated | 104

BASELINE CHARACTERISTICS:
Population: Full analysis set, defined as enrolled participants who received at least 1 dose of darbepoetin alfa or any other erythropoiesis-stimulating agent (ESA) before the end of study.
Arm/Group | Darbepoetin Alfa or Other ESA
Number analyzed (Participants) | 1158
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 691
  Male | 467
Fatigue-Visual Analog Scale (VAS) Score [Mean (Standard Deviation); unit: units on a scale] — The fatigue VAS is a 100-point scale where fatigue-levels are rated from 0 (least fatigue) to 100 (worst possible fatigue). Baseline VAS data were available for 1109 participants.
  units on a scale | 51.2 (22.6)
Functional Assessment of Cancer Therapy-Fatigue (FACT-F) score [Mean (Standard Deviation); unit: units on a scale] — The FACT-F subscale consists of 13 fatigue-related items that are a subset of the Functional Assessment of Cancer Therapy - Anaemia (FACT-An) questionnaire. Participants indicate how they feel in response to 13 statements on a scale from 0 for "Not at all" to 4 for "Very much". Total scores for the FACT-F subscale range from 0 to 52; the higher the score the better the quality of life. Baseline data were available for 1109 participants.
  units on a scale | 28.4 (10.5)
Hemoglobin level [Mean (Standard Deviation); unit: g/dL] — Baseline hemoglobin levels were available for 1133 participants.
  g/dL | 9.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving Darbepoetin Alfa With Improvement in Patient Perceived Fatigue (PPF) and Increase in Hemoglobin ≥ 1 g/dL
Description: Improvement in PPF was defined as improvement at Week 9 in Functional Assessment of Cancer Therapy-Fatigue (FACT-F) score of ≥ 3.5 points from Baseline (the minimally important difference [MID]), and an increase in hemoglobin was defined as ≥ 1 g/dL increase from Baseline. The FACT-F MID was determined by the mean FACT-F change score (between Baseline and Week 9) for participants who had an improvement in the fatigue visual analog scale (VAS) score of 5 ± 3 points. The FACT-F subscale consists of 13 fatigue-related items that are a subset of the Functional Assessment of Cancer Therapy - Anaemia (FACT-An) questionnaire. Participants indicate how they feel in response to 13 statements on a scale from 0 for "Not at all" to 4 for "Very much". Total scores for the FACT-F subscale range from 0 to 52; the higher the score the better the quality of life. The fatigue-VAS is a 100-point scale, where fatigue-levels are rated from 0 (least fatigue) to 100 (worst possible fatigue).
Time Frame: Baseline to Week 9 (Treatment Day 57). Due to the observational nature of the study and variation in ESA dosing schedules, assessments closest to day 57 and within Days 43 to 70 (inclusive) were used to calculate the Week 9 visit results.
Population: The Primary analysis set consists of enrolled participants who received at least 1 dose of darbepoetin alfa, have baseline assessments for each of Hemoglobin, FACT-F subscale and VAS, and analyzable post-baseline assessments for each of Hemoglobin, FACT-F subscale, and VAS at Week 9.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Darbepoetin Alfa: Participants receiving systemic chemotherapy for solid tumors who also received darbepoetin alfa (Aranesp®) to treat symptomatic anemia according to routine institutional practice.
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 510
percentage of participants | 31.8 [27.7 to 35.8]

2. Secondary Outcome: Percentage of Participants by Tumor Type With Improvement in Patient Perceived Fatigue (PPF) and Increase in Hemoglobin ≥ 1 g/dL
Description: as for outcome 1
Time Frame: Baseline to Week 9
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 510
percentage of participants
  Breast cancer (N=152) | 38.8 [31.1 to 46.6]
  Prostate cancer (N=39) | 28.2 [14.1 to 42.3]
  Small cell lung cancer (N=12) | 16.7 [0.0 to 37.8]
  Non-small cell lung cancer (N=70) | 28.6 [18.0 to 39.2]
  Colorectal cancer (N=71) | 31.0 [20.2 to 41.7]
  Ovarian cancer (N=79) | 38.0 [27.3 to 48.7]
  Bladder cancer (N=16) | 0.0 [NA to NA] — Confidence interval could not be calculated since there were no participants with both PPF improvement and hemoglobin increase.
  Endometrial cancer (N=12) | 8.3 [0.0 to 24.0]
  Renal cancer (N=10) | 10.0 [0.0 to 28.6]
  Pancreatic cancer (N=31) | 35.5 [18.6 to 52.3]
  Esophogeal cancer (N=3) | 33.3 [0.0 to 86.7]
  Gastric cancer (N=15) | 26.7 [4.3 to 49.0]

3. Secondary Outcome: Mean Change From Baseline in FACT-F Score for Participants With a VAS Improvement of 5 ± 3 Points
Description: The FACT-F subscale consists of 13 fatigue-related items (statements) that are a subset of the Functional Assessment of Cancer Therapy - Anaemia (FACT-An) questionnaire. Participants are asked to indicate how they feel in response to each of the 13 statements on a scale from 0 for "Not at all" to 4 for "Very much". Total scores for the FACT-F subscale can range from 0 to 52; the higher the score the better the quality of life. A positive change (>0) from baseline score constitutes an improvement in fatigue between Baseline and Week 9. The fatigue-visual analog scale (VAS) is a 100-point scale where fatigue-levels are rated from 0 (least fatigue) to 100 (worst possible fatigue).
Time Frame: Baseline and Week 9
Population: Primary analysis set participants with a fatigue VAS score improvement at Week 9 of 5 ± 3 points from Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 44
units on a scale | 3.5 (5.5)

4. Secondary Outcome: Time to First Increase in Hemoglobin
Description: Time from Baseline to first increase in hemoglobin of ≥ 1 g/dL
Time Frame: From Baseline until Week 9
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 510
days | 36.5 [30.0 to 43.0]

5. Secondary Outcome: Percentage of Participants With Improvement in Patient-perceived Fatigue (PPF) at Any Time
Description: The percentage of participants with iimprovement in PPF at any time from Day 2 until the end-of-study assessment (Week 13). Improvement in PPF was defined as improvement in Functional Assessment of Cancer Therapy-Fatigue (FACT-F) score of ≥ 3.5 points from Baseline (the minimally important difference [MID]). The FACT-F MID was determined by the mean FACT-F change score (between Baseline and Week 9) for participants who had an improvement in the fatigue visual analog scale (VAS) score of 5 ± 3 points. The FACT-F subscale consists of 13 fatigue-related items that are a subset of the FACT-An questionnaire. Participants indicate how they feel in response to 13 statements on a scale from 0 for "Not at all" to 4 for "Very much". Total scores for the FACT-F subscale range from 0 to 52; the higher the score the better the quality of life. The fatigue-VAS is a 100-point scale, where fatigue-levels are rated from 0 (least fatigue) to 100 (worst possible fatigue).
Time Frame: From Baseline to Week 13
Population: Primary analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 510
percentage of participants | 70.0

6. Secondary Outcome: Percentage of Participants With Increase in Hemoglobin ≥ 1 g/dL at Any Time
Description: The percentage of participants with increase in hemoglobin (≥ 1 g/dL) at any time from Day 2 until the end-of-study assessment (Week 13).
Time Frame: From Baseline to Week 13
Population: Primary analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 510
percentage of participants | 75.7

ADVERSE EVENTS:
Time Frame: Up to 28 days after a participant's last dose date, capped at 17 weeks
Description: Only adverse drug reactions to Amgen products were collected in this study. The table of Other Adverse Events summarizes non-serious occurrences of adverse drug reactions.
Arm/Group | Darbepoetin Alfa or Other ESA
Serious Adverse Events (participants affected / at risk) | 2/1158
Other Adverse Events (participants affected / at risk) | 8/1158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa or Other ESA (N=1158)
Cardiac arrest (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa or Other ESA (N=1158)
Thrombocytosis (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cystoid macular oedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Injection site pain (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.